CLINICAL TRIAL: NCT05108896
Title: Aspiration in Acute Respiratory Failure Survivors
Brief Title: Aspiration in Acute Respiratory Failure Survivors 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-3873; R01NR019989 (NIH)
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Dysphagia; Aspiration
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Multi-center prospective single cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspiration in Acute Respiratory Failure Survivors (Other): All participants will receive a tracheal ultrasound within 72 hours prior to extubation, collection of demographic and hospital clinical information, administration of 3 screening tests (study defined algorithm test, 3-ounce water swallow test, TOR-BSST) addressing swallowing function within 24 hours post-extubation, and a fiberoptic endoscopic examination of swallowing (FEES) exam.
  Interventions: Diagnostic Test: 3-Screenings Protocol; Diagnostic Test: FEES; Diagnostic Test: Tracheal Ultrasound

INTERVENTIONS:
Diagnostic Test: 3-Screenings Protocol — The 3-Screenings Protocol is a modified bedside swallow exam (BSE) consisting of a study developed five-item decision tree algorithm including voice quality assessment and a 2-ounce water consistency assessment, the Yale Swallow Test, with a scored 3-ounce Water Swallow Test (3-WST), and the Toronto Bedside Swallowing Screening Test (TOR-BSST).
  Other Names: Modified bedside swallow exam (BSE); Three Screening Tests
Diagnostic Test: FEES — A thin, flexible endoscope designed for assessment of laryngeal structures is passed through the nose to the oropharynx, visualizing the laryngeal structures, and the base of tongue and the pharynx. If needed 4% topical lidocaine and/or oxymetazoline (Afrin) will be administered. Swallowing will then be evaluated directly with six food boluses of 5 ml each. All patients will be allowed to swallow spontaneously without a verbal command to swallow. Video of the examinations will be recorded and presence of dysphagia will be designated independently by 3 different observers (one pulmonary physician and two speech language pathologists (SLPs)). This procedure will take 5-10 minutes. The camera will then be removed.
  Other Names: Fiberoptic Endoscopic Evaluation of Swallowing
Diagnostic Test: Tracheal Ultrasound — Ultrasound imaging of the trachea, measuring tracheal diameter and endotracheal tube (ETT) size ratio within 72 hours prior to extubation

SUMMARY:
The purpose of this study is to learn more about problems with swallowing that could develop in patients who are very sick and need a machine to help them breathe.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about problems with swallowing that could develop in patients who are very sick and need a machine to help them breathe. Patients are asked to be in this study because they had problems breathing on their own and therefore needed the help of a machine called a ventilator. In order for this ventilator to push air into the lungs, patients need a tube placed in the throat called an endotracheal tube. The process of placing this endotracheal tube was called intubation. The tube has now been removed, which is a process called extubation. Sometimes, people who have had endotracheal tubes can have difficulty swallowing food and liquids for a period of time. This disease is called post-extubation dysphagia (PED). PED is a serious condition and may result in food or liquid going from the mouth into the lungs. This could cause further lung problems. Given this risk, doctors sometimes suggest that patients with PED either avoid eating or drinking, or get a feeding tube. Currently, nobody knows how often patients develop PED, why they develop it, or the best method to detect it. Standard care involves clinicians making educated guesses. This study looks to determine if watching the patient swallow, both with and without a small camera, is an accurate method for detecting PED.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to an ICU.
2. Mechanical ventilation with an endotracheal tube for greater than 48 hours.

Exclusion Criteria:

1. Likely persistent contraindications to enteral/oral nutrition administration.
2. Pre-existing history of dysphagia or aspiration.
3. Pre-existing or acute primary central or peripheral neuromuscular disorder.
4. Presence of a chronic tracheostomy (present prior to ICU admission).
5. Pre-existing head and neck cancer or surgery.
6. Coagulopathy resulting in uncontrolled nasal or pharyngeal bleeding.
7. Delirium for more than 96 hours after extubation as assessed by Confusion Assessment Method (CAM-ICU).
8. Extubated for greater than 96 hours.
9. Inability to obtain informed consent from patient or an appropriate surrogate.
10. Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 855 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing aspiration on the FEES with any of the feeding consistencies | from extubation day 1 through hospital discharge, expected to be within 28 days
  Aspiration (PAS score of ≥6) on the FEES with any of the feeding consistencies. A PAS score of ≥ 6 includes patients with both silent and non-silent aspiration. Using a PAS cutoff score of ≥6 on FEES, patients will be stratified by aspiration on any of the five consistencies.

SECONDARY OUTCOMES:
Percentage of participants experiencing non-silent aspiration | from extubation day 1 through hospital discharge, expected to be within 28 days
  We will stratify patients who aspirate into non-silent (PA = 6- 7) and silent (PAS=8) aspiration, and also determine maximum PAS scores across bolus and consistency types. Aspiration (PAS score of ≥6) on the FEES with any of the feeding consistencies. A PAS score of ≥ 6 includes patients with both silent and non-silent aspiration. Using a PAS cutoff score of ≥6 on FEES, patients will be stratified by aspiration on any of the five consistencies. We will also determine the maximum PAS scores across bolus and consistency types.
Percentage of participants experiencing silent aspiration | from extubation day 1 through hospital discharge, expected to be within 28 days
  We will stratify patients who aspirate into non-silent (PA = 6- 7) and silent (PAS=8) aspiration, and also determine maximum PAS scores across bolus and consistency types. Aspiration (PAS score of ≥6) on the FEES with any of the feeding consistencies. A PAS score of ≥ 6 includes patients with both silent and non-silent aspiration. Using a PAS cutoff score of ≥6 on FEES, patients will be stratified by aspiration on any of the five consistencies. We will also determine the maximum PAS scores across bolus and consistency types.
Percentage of participants experiencing post-extubation clinical laryngeal edema | Within 24 hours after extubation
  We will define laryngeal edema as upper-airway obstruction within 24 hours after extubation. Minor laryngeal edema will be defined as stridor associated with a respiratory distress defined as a prolonged inspiratory phase and the presence of edema on FEES examination. Major laryngeal edema will defined as severe respiratory distress needing tracheal reintubation secondary to upper-airway obstruction that was visualized during the FEES examination
Duration of mechanical ventilation | from intubation and receipt of mechanical ventilation through extubation, expected to be within 2-14 days on average
  We will also collect the overall length of mechanical ventilation in days
Duration required for liberation from mechanical ventilation | from intubation and receipt of mechanical ventilation through extubation, expected to be within 2-14 days on average
  We will also collect the overall length of the liberation process from mechanical ventilation in days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- United States (5):
  - Stanford Univerity, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University, Boston, Massachusetts

REFERENCES:
- [Background] Kempker JA, Abril MK, Chen Y, Kramer MR, Waller LA, Martin GS. The Epidemiology of Respiratory Failure in the United States 2002-2017: A Serial Cross-Sectional Study. Crit Care Explor. 2020 Jun 10;2(6):e0128. doi: 10.1097/CCE.0000000000000128. eCollection 2020 Jun. PMID 32695994
- [Background] Wunsch H, Linde-Zwirble WT, Angus DC, Hartman ME, Milbrandt EB, Kahn JM. The epidemiology of mechanical ventilation use in the United States. Crit Care Med. 2010 Oct;38(10):1947-53. doi: 10.1097/CCM.0b013e3181ef4460. PMID 20639743
- [Background] Barker J, Martino R, Reichardt B, Hickey EJ, Ralph-Edwards A. Incidence and impact of dysphagia in patients receiving prolonged endotracheal intubation after cardiac surgery. Can J Surg. 2009 Apr;52(2):119-24. PMID 19399206
- [Background] El Solh A, Okada M, Bhat A, Pietrantoni C. Swallowing disorders post orotracheal intubation in the elderly. Intensive Care Med. 2003 Sep;29(9):1451-5. doi: 10.1007/s00134-003-1870-4. Epub 2003 Aug 2. PMID 12904855
- [Background] Macht M, White SD, Moss M. Swallowing dysfunction after critical illness. Chest. 2014 Dec;146(6):1681-1689. doi: 10.1378/chest.14-1133. PMID 25451355
- [Background] Macht M, Wimbish T, Bodine C, Moss M. ICU-acquired swallowing disorders. Crit Care Med. 2013 Oct;41(10):2396-405. doi: 10.1097/CCM.0b013e31829caf33. PMID 23939361
- [Background] Skoretz SA, Flowers HL, Martino R. The incidence of dysphagia following endotracheal intubation: a systematic review. Chest. 2010 Mar;137(3):665-73. doi: 10.1378/chest.09-1823. PMID 20202948
- [Background] Moss M, White SD, Warner H, Dvorkin D, Fink D, Gomez-Taborda S, Higgins C, Krisciunas GP, Levitt JE, McKeehan J, McNally E, Rubio A, Scheel R, Siner JM, Vojnik R, Langmore SE. Development of an Accurate Bedside Swallowing Evaluation Decision Tree Algorithm for Detecting Aspiration in Acute Respiratory Failure Survivors. Chest. 2020 Nov;158(5):1923-1933. doi: 10.1016/j.chest.2020.07.051. Epub 2020 Jul 25. PMID 32721404
- [Background] Borders JC, Fink D, Levitt JE, McKeehan J, McNally E, Rubio A, Scheel R, Siner JM, Taborda SG, Vojnik R, Warner H, White SD, Langmore SE, Moss M, Krisciunas GP. Relationship Between Laryngeal Sensation, Length of Intubation, and Aspiration in Patients with Acute Respiratory Failure. Dysphagia. 2019 Aug;34(4):521-528. doi: 10.1007/s00455-019-09980-1. Epub 2019 Jan 29. PMID 30694412
- [Background] Krisciunas GP, Langmore SE, Gomez-Taborda S, Fink D, Levitt JE, McKeehan J, McNally E, Scheel R, Rubio AC, Siner JM, Vojnik R, Warner H, White SD, Moss M. The Association Between Endotracheal Tube Size and Aspiration (During Flexible Endoscopic Evaluation of Swallowing) in Acute Respiratory Failure Survivors. Crit Care Med. 2020 Nov;48(11):1604-1611. doi: 10.1097/CCM.0000000000004554. PMID 32804785
- [Background] DePippo KL, Holas MA, Reding MJ. Validation of the 3-oz water swallow test for aspiration following stroke. Arch Neurol. 1992 Dec;49(12):1259-61. doi: 10.1001/archneur.1992.00530360057018. PMID 1449405
- [Background] Martino R, Silver F, Teasell R, Bayley M, Nicholson G, Streiner DL, Diamant NE. The Toronto Bedside Swallowing Screening Test (TOR-BSST): development and validation of a dysphagia screening tool for patients with stroke. Stroke. 2009 Feb;40(2):555-61. doi: 10.1161/STROKEAHA.107.510370. Epub 2008 Dec 12. PMID 19074483
- [Background] Suiter DM, Leder SB. Clinical utility of the 3-ounce water swallow test. Dysphagia. 2008 Sep;23(3):244-50. doi: 10.1007/s00455-007-9127-y. Epub 2007 Dec 4. PMID 18058175
- [Background] Suiter DM, Sloggy J, Leder SB. Validation of the Yale Swallow Protocol: a prospective double-blinded videofluoroscopic study. Dysphagia. 2014 Apr;29(2):199-203. doi: 10.1007/s00455-013-9488-3. Epub 2013 Sep 12. PMID 24026519
- [Background] Langmore SE. Role of flexible laryngoscopy for evaluating aspiration. Ann Otol Rhinol Laryngol. 1998 May;107(5 Pt 1):446. doi: 10.1177/000348949810700516. No abstract available. PMID 9596227
- [Background] Sinha P, Calfee CS, Cherian S, Brealey D, Cutler S, King C, Killick C, Richards O, Cheema Y, Bailey C, Reddy K, Delucchi KL, Shankar-Hari M, Gordon AC, Shyamsundar M, O'Kane CM, McAuley DF, Szakmany T. Prevalence of phenotypes of acute respiratory distress syndrome in critically ill patients with COVID-19: a prospective observational study. Lancet Respir Med. 2020 Dec;8(12):1209-1218. doi: 10.1016/S2213-2600(20)30366-0. Epub 2020 Aug 27. PMID 32861275
- [Background] Sinha P, Calfee CS. Phenotypes in acute respiratory distress syndrome: moving towards precision medicine. Curr Opin Crit Care. 2019 Feb;25(1):12-20. doi: 10.1097/MCC.0000000000000571. PMID 30531367
- [Background] Sinha P, Calfee CS. Peeking under the Hood of Acute Respiratory Distress Syndrome Phenotypes: Deeper Insights into Biological Heterogeneity. Am J Respir Crit Care Med. 2019 Jul 1;200(1):4-6. doi: 10.1164/rccm.201901-0195ED. No abstract available. PMID 30753791
- [Background] Reilly JP, Calfee CS, Christie JD. Acute Respiratory Distress Syndrome Phenotypes. Semin Respir Crit Care Med. 2019 Feb;40(1):19-30. doi: 10.1055/s-0039-1684049. Epub 2019 May 6. PMID 31060085
- [Background] Lakhal K, Delplace X, Cottier JP, Tranquart F, Sauvagnac X, Mercier C, Fusciardi J, Laffon M. The feasibility of ultrasound to assess subglottic diameter. Anesth Analg. 2007 Mar;104(3):611-4. doi: 10.1213/01.ane.0000260136.53694.fe. PMID 17312218
- [Background] Gollu G, Onat Bermede A, Khanmammadov F, Ates U, Genc S, Selvi Can O, Fitoz S, Alanoglu Z, Yagmurlu A. Use of ultrasonography as a noninvasive decisive tool to determine the accurate endotracheal tube size in anesthetized children. Arch Argent Pediatr. 2018 Jun 1;116(3):172-178. doi: 10.5546/aap.2018.eng.172. English, Spanish. PMID 29756700
- [Background] Maloney JP, Halbower AC, Fouty BF, Fagan KA, Balasubramaniam V, Pike AW, Fennessey PV, Moss M. Systemic absorption of food dye in patients with sepsis. N Engl J Med. 2000 Oct 5;343(14):1047-8. doi: 10.1056/NEJM200010053431416. No abstract available. PMID 11023403
- [Background] Langmore SE. Efficacy of behavioral treatment for oropharyngeal dysphagia. Dysphagia. 1995 Fall;10(4):259-62. doi: 10.1007/BF00431419. PMID 7493507
- [Background] Langmore SE. Dysphagia in neurologic patients in the intensive care unit. Semin Neurol. 1996 Dec;16(4):329-40. doi: 10.1055/s-2008-1040991. No abstract available. PMID 9112312
- [Background] Langmore SE. Laryngeal sensation: a touchy subject. Dysphagia. 1998 Spring;13(2):93-4. No abstract available. PMID 9513303
- [Background] Langmore SE. Issues in the management of dysphagia. Folia Phoniatr Logop. 1999 Jul-Oct;51(4-5):220-30. doi: 10.1159/000021499. PMID 10450028
- [Background] Langmore SE. An important tool for measuring quality of life. Dysphagia. 2000 Summer;15(3):134-5. doi: 10.1007/s004550010014. No abstract available. PMID 10839825
- [Background] Langmore SE. Evaluation of oropharyngeal dysphagia: which diagnostic tool is superior? Curr Opin Otolaryngol Head Neck Surg. 2003 Dec;11(6):485-9. doi: 10.1097/00020840-200312000-00014. PMID 14631184
- [Background] Langmore SE, Grillone G, Elackattu A, Walsh M. Disorders of swallowing: palliative care. Otolaryngol Clin North Am. 2009 Feb;42(1):87-105, ix. doi: 10.1016/j.otc.2008.09.005. PMID 19134493
- [Background] Langmore SE, Kasarskis EJ, Manca ML, Olney RK. Enteral tube feeding for amyotrophic lateral sclerosis/motor neuron disease. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD004030. doi: 10.1002/14651858.CD004030.pub2. PMID 17054194
- [Background] Langmore SE, Lehman ME. Physiologic deficits in the orofacial system underlying dysarthria in amyotrophic lateral sclerosis. J Speech Hear Res. 1994 Feb;37(1):28-37. doi: 10.1044/jshr.3701.28. PMID 8170127
- [Background] Langmore SE, Miller RM. Behavioral treatment for adults with oropharyngeal dysphagia. Arch Phys Med Rehabil. 1994 Oct;75(10):1154-60. doi: 10.1016/0003-9993(94)90094-9. PMID 7944924
- [Background] Langmore SE, Olney RK, Lomen-Hoerth C, Miller BL. Dysphagia in patients with frontotemporal lobar dementia. Arch Neurol. 2007 Jan;64(1):58-62. doi: 10.1001/archneur.64.1.58. PMID 17210809
- [Background] Langmore SE, Schatz K, Olsen N. Fiberoptic endoscopic examination of swallowing safety: a new procedure. Dysphagia. 1988;2(4):216-9. doi: 10.1007/BF02414429. No abstract available. PMID 3251697
- [Background] Langmore SE, Schatz K, Olson N. Endoscopic and videofluoroscopic evaluations of swallowing and aspiration. Ann Otol Rhinol Laryngol. 1991 Aug;100(8):678-81. doi: 10.1177/000348949110000815. PMID 1872520
- [Background] Langmore SE, Skarupski KA, Park PS, Fries BE. Predictors of aspiration pneumonia in nursing home residents. Dysphagia. 2002 Fall;17(4):298-307. doi: 10.1007/s00455-002-0072-5. PMID 12355145
- [Background] Langmore SE, Terpenning MS, Schork A, Chen Y, Murray JT, Lopatin D, Loesche WJ. Predictors of aspiration pneumonia: how important is dysphagia? Dysphagia. 1998 Spring;13(2):69-81. doi: 10.1007/PL00009559. PMID 9513300
- [Background] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Background] Adhikari NKJ, McAndrews MP, Tansey CM, Matte A, Pinto R, Cheung AM, Diaz-Granados N, Barr A, Herridge MS. Self-reported symptoms of depression and memory dysfunction in survivors of ARDS. Chest. 2009 Mar;135(3):678-687. doi: 10.1378/chest.08-0974. PMID 19265087
- [Background] Desai SV, Law TJ, Needham DM. Long-term complications of critical care. Crit Care Med. 2011 Feb;39(2):371-9. doi: 10.1097/CCM.0b013e3181fd66e5. PMID 20959786
- [Background] Griffiths RD, Jones C. Recovery from intensive care. BMJ. 1999 Aug 14;319(7207):427-9. doi: 10.1136/bmj.319.7207.427. No abstract available. PMID 10445926
- [Background] Herridge MS. Recovery and long-term outcome in acute respiratory distress syndrome. Crit Care Clin. 2011 Jul;27(3):685-704. doi: 10.1016/j.ccc.2011.04.003. PMID 21742223
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Hopkins RO, Weaver LK, Collingridge D, Parkinson RB, Chan KJ, Orme JF Jr. Two-year cognitive, emotional, and quality-of-life outcomes in acute respiratory distress syndrome. Am J Respir Crit Care Med. 2005 Feb 15;171(4):340-7. doi: 10.1164/rccm.200406-763OC. Epub 2004 Nov 12. PMID 15542793
- [Background] Daniels SK, Anderson JA, Willson PC. Valid items for screening dysphagia risk in patients with stroke: a systematic review. Stroke. 2012 Mar;43(3):892-7. doi: 10.1161/STROKEAHA.111.640946. Epub 2012 Feb 2. PMID 22308250
- [Background] Schepp SK, Tirschwell DL, Miller RM, Longstreth WT Jr. Swallowing screens after acute stroke: a systematic review. Stroke. 2012 Mar;43(3):869-71. doi: 10.1161/STROKEAHA.111.638254. Epub 2011 Dec 8. PMID 22156697
- [Background] Scott A, Perry A, Bench J. A study of interrater reliability when using videofluoroscopy as an assessment of swallowing. Dysphagia. 1998 Fall;13(4):223-7. doi: 10.1007/PL00009576. PMID 9716754
- [Background] Seymour CW, Kennedy JN, Wang S, Chang CH, Elliott CF, Xu Z, Berry S, Clermont G, Cooper G, Gomez H, Huang DT, Kellum JA, Mi Q, Opal SM, Talisa V, van der Poll T, Visweswaran S, Vodovotz Y, Weiss JC, Yealy DM, Yende S, Angus DC. Derivation, Validation, and Potential Treatment Implications of Novel Clinical Phenotypes for Sepsis. JAMA. 2019 May 28;321(20):2003-2017. doi: 10.1001/jama.2019.5791. PMID 31104070
- [Background] Bours GJ, Speyer R, Lemmens J, Limburg M, de Wit R. Bedside screening tests vs. videofluoroscopy or fibreoptic endoscopic evaluation of swallowing to detect dysphagia in patients with neurological disorders: systematic review. J Adv Nurs. 2009 Mar;65(3):477-93. doi: 10.1111/j.1365-2648.2008.04915.x. PMID 19222645
- [Background] Carnaby G, Hankey GJ, Pizzi J. Behavioural intervention for dysphagia in acute stroke: a randomised controlled trial. Lancet Neurol. 2006 Jan;5(1):31-7. doi: 10.1016/S1474-4422(05)70252-0. PMID 16361020
- [Background] Carnaby-Mann GD, Crary MA. McNeill dysphagia therapy program: a case-control study. Arch Phys Med Rehabil. 2010 May;91(5):743-9. doi: 10.1016/j.apmr.2010.01.013. PMID 20434612
- [Background] DePippo KL, Holas MA, Reding MJ, Mandel FS, Lesser ML. Dysphagia therapy following stroke: a controlled trial. Neurology. 1994 Sep;44(9):1655-60. doi: 10.1212/wnl.44.9.1655. PMID 7936292
- [Background] Duarte VM, Chhetri DK, Liu YF, Erman AA, Wang MB. Swallow preservation exercises during chemoradiation therapy maintains swallow function. Otolaryngol Head Neck Surg. 2013 Dec;149(6):878-84. doi: 10.1177/0194599813502310. Epub 2013 Aug 27. PMID 23981953
- [Background] Logemann JA. Treatment of oral and pharyngeal dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):803-16, ix. doi: 10.1016/j.pmr.2008.06.003. PMID 18940642
- [Background] Logemann JA, Gensler G, Robbins J, Lindblad AS, Brandt D, Hind JA, Kosek S, Dikeman K, Kazandjian M, Gramigna GD, Lundy D, McGarvey-Toler S, Miller Gardner PJ. A randomized study of three interventions for aspiration of thin liquids in patients with dementia or Parkinson's disease. J Speech Lang Hear Res. 2008 Feb;51(1):173-83. doi: 10.1044/1092-4388(2008/013). PMID 18230864
- [Background] Logemann JA, Pauloski BR, Rademaker AW, Lazarus CL, Gaziano J, Stachowiak L, Newman L, MacCracken E, Santa D, Mittal B. Swallowing disorders in the first year after radiation and chemoradiation. Head Neck. 2008 Feb;30(2):148-58. doi: 10.1002/hed.20672. PMID 17786992
- [Background] Logemann JA, Rademaker A, Pauloski BR, Antinoja J, Bacon M, Bernstein M, Gaziano J, Grande B, Kelchner L, Kelly A, Klaben B, Lundy D, Newman L, Santa D, Stachowiak L, Stangl-McBreen C, Atkinson C, Bassani H, Czapla M, Farquharson J, Larsen K, Lewis V, Logan H, Nitschke T, Veis S. What information do clinicians use in recommending oral versus nonoral feeding in oropharyngeal dysphagic patients? Dysphagia. 2008 Dec;23(4):378-84. doi: 10.1007/s00455-008-9152-5. Epub 2008 Aug 1. PMID 18670808
- [Background] Logemann JA, Rademaker A, Pauloski BR, Kelly A, Stangl-McBreen C, Antinoja J, Grande B, Farquharson J, Kern M, Easterling C, Shaker R. A randomized study comparing the Shaker exercise with traditional therapy: a preliminary study. Dysphagia. 2009 Dec;24(4):403-11. doi: 10.1007/s00455-009-9217-0. Epub 2009 May 27. PMID 19472007
- [Background] Robbins J, Gensler G, Hind J, Logemann JA, Lindblad AS, Brandt D, Baum H, Lilienfeld D, Kosek S, Lundy D, Dikeman K, Kazandjian M, Gramigna GD, McGarvey-Toler S, Miller Gardner PJ. Comparison of 2 interventions for liquid aspiration on pneumonia incidence: a randomized trial. Ann Intern Med. 2008 Apr 1;148(7):509-18. doi: 10.7326/0003-4819-148-7-200804010-00007. PMID 18378947
- [Background] Speyer R, Baijens L, Heijnen M, Zwijnenberg I. Effects of therapy in oropharyngeal dysphagia by speech and language therapists: a systematic review. Dysphagia. 2010 Mar;25(1):40-65. doi: 10.1007/s00455-009-9239-7. Epub 2009 Sep 17. PMID 19760458
- [Background] Brodsky MB, De I, Chilukuri K, Huang M, Palmer JB, Needham DM. Coordination of Pharyngeal and Laryngeal Swallowing Events During Single Liquid Swallows After Oral Endotracheal Intubation for Patients with Acute Respiratory Distress Syndrome. Dysphagia. 2018 Dec;33(6):768-777. doi: 10.1007/s00455-018-9901-z. Epub 2018 Apr 30. PMID 29713897
- [Background] Francois B, Bellissant E, Gissot V, Desachy A, Normand S, Boulain T, Brenet O, Preux PM, Vignon P; Association des Reanimateurs du Centre-Ouest (ARCO). 12-h pretreatment with methylprednisolone versus placebo for prevention of postextubation laryngeal oedema: a randomised double-blind trial. Lancet. 2007 Mar 31;369(9567):1083-9. doi: 10.1016/S0140-6736(07)60526-1. PMID 17398307
- [Background] Lynch YT, Clark BJ, Macht M, White SD, Taylor H, Wimbish T, Moss M. The accuracy of the bedside swallowing evaluation for detecting aspiration in survivors of acute respiratory failure. J Crit Care. 2017 Jun;39:143-148. doi: 10.1016/j.jcrc.2017.02.013. Epub 2017 Feb 15. PMID 28259057
- [Background] Gupta B, Gupta L. Significance of the outer diameter of an endotracheal tube: a lesser-known parameter. Korean J Anesthesiol. 2019 Feb;72(1):72-73. doi: 10.4097/kja.d.18.00056. Epub 2018 May 30. No abstract available. PMID 29843505
- [Background] Farrow S, Farrow C, Soni N. Size matters: choosing the right tracheal tube. Anaesthesia. 2012 Aug;67(8):815-9. doi: 10.1111/j.1365-2044.2012.07250.x. No abstract available. PMID 22775368
- [Background] Bae JY, Byon HJ, Han SS, Kim HS, Kim JT. Usefulness of ultrasound for selecting a correctly sized uncuffed tracheal tube for paediatric patients. Anaesthesia. 2011 Nov;66(11):994-8. doi: 10.1111/j.1365-2044.2011.06900.x. Epub 2011 Sep 20. PMID 21933159
- [Background] Levine ME. The four conservation principles of nursing. Nurs Forum. 1967;6(1):45-59. doi: 10.1111/j.1744-6198.1967.tb01297.x. No abstract available. PMID 5180875
- [Background] Levine ME. The conservation principles: a retrospective. Nurs Sci Q. 1996 Spring;9(1):38-41. doi: 10.1177/089431849600900110. No abstract available. PMID 8710302
- [Background] Goldman L, Weinberg M, Weisberg M, Olshen R, Cook EF, Sargent RK, Lamas GA, Dennis C, Wilson C, Deckelbaum L, Fineberg H, Stiratelli R. A computer-derived protocol to aid in the diagnosis of emergency room patients with acute chest pain. N Engl J Med. 1982 Sep 2;307(10):588-96. doi: 10.1056/NEJM198209023071004. PMID 7110205
- [Background] Hoffman JR, Mower WR, Wolfson AB, Todd KH, Zucker MI. Validity of a set of clinical criteria to rule out injury to the cervical spine in patients with blunt trauma. National Emergency X-Radiography Utilization Study Group. N Engl J Med. 2000 Jul 13;343(2):94-9. doi: 10.1056/NEJM200007133430203. PMID 10891516
- [Background] Macht M, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Postextubation dysphagia is persistent and associated with poor outcomes in survivors of critical illness. Crit Care. 2011;15(5):R231. doi: 10.1186/cc10472. Epub 2011 Sep 29. PMID 21958475
- [Background] Macht M, Wimbish T, Clark BJ, Benson AB, Burnham EL, Williams A, Moss M. Diagnosis and treatment of post-extubation dysphagia: results from a national survey. J Crit Care. 2012 Dec;27(6):578-86. doi: 10.1016/j.jcrc.2012.07.016. Epub 2012 Oct 18. PMID 23084136
- [Background] Brown AW, Malec JF, McClelland RL, Diehl NN, Englander J, Cifu DX. Clinical elements that predict outcome after traumatic brain injury: a prospective multicenter recursive partitioning (decision-tree) analysis. J Neurotrauma. 2005 Oct;22(10):1040-51. doi: 10.1089/neu.2005.22.1040. PMID 16238482
- [Background] Seheult JN, Anto VP, Farhat N, Stram MN, Spinella PC, Alarcon L, Sperry J, Triulzi DJ, Yazer MH. Application of a recursive partitioning decision tree algorithm for the prediction of massive transfusion in civilian trauma: the MTPitt prediction tool. Transfusion. 2019 Mar;59(3):953-964. doi: 10.1111/trf.15078. Epub 2018 Dec 12. PMID 30548461
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Bryant LR, Trinkle JK, Mobin-Uddin K, Baker J, Griffen WO Jr. Bacterial colonization profile with tracheal intubation and mechanical ventilation. Arch Surg. 1972 May;104(5):647-51. doi: 10.1001/archsurg.1972.04180050023006. No abstract available. PMID 4402112
- [Background] Johanson WG, Pierce AK, Sanford JP. Changing pharyngeal bacterial flora of hospitalized patients. Emergence of gram-negative bacilli. N Engl J Med. 1969 Nov 20;281(21):1137-40. doi: 10.1056/NEJM196911202812101. No abstract available. PMID 4899868
- [Background] Ely EW, Siegel MD, Inouye SK. Delirium in the intensive care unit: an under-recognized syndrome of organ dysfunction. Semin Respir Crit Care Med. 2001;22(2):115-26. doi: 10.1055/s-2001-13826. PMID 16088667
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Vazquez R, Gheorghe C, Ramos F, Dadu R, Amoateng-Adjepong Y, Manthous CA. Gurgling breath sounds may predict hospital-acquired pneumonia. Chest. 2010 Aug;138(2):284-8. doi: 10.1378/chest.09-2713. Epub 2010 Mar 26. PMID 20348197
- [Background] Martino R, Maki E, Diamant N. Identification of dysphagia using the Toronto Bedside Swallowing Screening Test (TOR-BSST(c)): are 10 teaspoons of water necessary? Int J Speech Lang Pathol. 2014 Jun;16(3):193-8. doi: 10.3109/17549507.2014.902995. PMID 24833425
- [Background] Pacheco-Castilho AC, de Martini Vanin G, Reichardt B, Miranda RPC, Norberto AMQ, Braga MC, Bueno TBC, Weber KT, Santos TEG, Leite JP, Dantas RO, Pontes-Neto OM, Martino R. Translation and Validation of the TOR-BSST(c) into Brazilian Portuguese for Adults with Stroke. Dysphagia. 2021 Aug;36(4):533-540. doi: 10.1007/s00455-020-10167-2. Epub 2020 Aug 6. PMID 32766936
- [Background] Cho HM, Yoo B. Rheological characteristics of cold thickened beverages containing xanthan gum-based food thickeners used for dysphagia diets. J Acad Nutr Diet. 2015 Jan;115(1):106-11. doi: 10.1016/j.jand.2014.08.028. Epub 2014 Nov 4. PMID 25441963
- [Background] Cichero JA, Lam P, Steele CM, Hanson B, Chen J, Dantas RO, Duivestein J, Kayashita J, Lecko C, Murray J, Pillay M, Riquelme L, Stanschus S. Development of International Terminology and Definitions for Texture-Modified Foods and Thickened Fluids Used in Dysphagia Management: The IDDSI Framework. Dysphagia. 2017 Apr;32(2):293-314. doi: 10.1007/s00455-016-9758-y. Epub 2016 Dec 2. PMID 27913916
- [Background] Park J, Yoo W, Yoo B. Standard Recipes for the Preparation of Thickened Barium Liquids Used in the Diagnosis of Dysphagia. Clin Nutr Res. 2019 Oct 25;8(4):265-271. doi: 10.7762/cnr.2019.8.4.265. eCollection 2019 Oct. PMID 31720252
- [Background] Seo CW, Yoo B. Steady and dynamic shear rheological properties of gum-based food thickeners used for diet modification of patients with dysphagia: effect of concentration. Dysphagia. 2013 Jun;28(2):205-11. doi: 10.1007/s00455-012-9433-x. Epub 2012 Nov 24. PMID 23179025
- [Background] Rosenbek JC, Robbins JA, Roecker EB, Coyle JL, Wood JL. A penetration-aspiration scale. Dysphagia. 1996 Spring;11(2):93-8. doi: 10.1007/BF00417897. PMID 8721066
- [Background] Colodny N. Interjudge and intrajudge reliabilities in fiberoptic endoscopic evaluation of swallowing (fees) using the penetration-aspiration scale: a replication study. Dysphagia. 2002 Fall;17(4):308-15. doi: 10.1007/s00455-002-0073-4. PMID 12355146
- [Background] Kelly AM, Leslie P, Beale T, Payten C, Drinnan MJ. Fibreoptic endoscopic evaluation of swallowing and videofluoroscopy: does examination type influence perception of pharyngeal residue severity? Clin Otolaryngol. 2006 Oct;31(5):425-32. doi: 10.1111/j.1749-4486.2006.01292.x. PMID 17014453
- [Background] Kelly AM, Drinnan MJ, Leslie P. Assessing penetration and aspiration: how do videofluoroscopy and fiberoptic endoscopic evaluation of swallowing compare? Laryngoscope. 2007 Oct;117(10):1723-7. doi: 10.1097/MLG.0b013e318123ee6a. PMID 17906496
- [Background] Leder SB, Acton LM, Lisitano HL, Murray JT. Fiberoptic endoscopic evaluation of swallowing (FEES) with and without blue-dyed food. Dysphagia. 2005 Spring;20(2):157-62. doi: 10.1007/s00455-005-0009-x. PMID 16172826
- [Background] Fife TA, Butler SG, Langmore SE, Lester S, Wright SC Jr, Kemp S, Grace-Martin K, Lintzenich CR. Use of topical nasal anesthesia during flexible endoscopic evaluation of swallowing in dysphagic patients. Ann Otol Rhinol Laryngol. 2015 Mar;124(3):206-11. doi: 10.1177/0003489414550153. Epub 2014 Sep 9. PMID 25204714
- [Background] Lester S, Langmore SE, Lintzenich CR, Wright SC, Grace-Martin K, Fife T, Butler SG. The effects of topical anesthetic on swallowing during nasoendoscopy. Laryngoscope. 2013 Jul;123(7):1704-8. doi: 10.1002/lary.23899. Epub 2013 Apr 2. PMID 23553259
- [Background] Sadek SA, De R, Scott A, White AP, Wilson PS, Carlin WV. The efficacy of topical anaesthesia in flexible nasendoscopy: a double-blind randomised controlled trial. Clin Otolaryngol Allied Sci. 2001 Feb;26(1):25-8. doi: 10.1046/j.1365-2273.2001.00400.x. PMID 11298162
- [Background] Sunkaraneni VS, Jones SE. Topical anaesthetic or vasoconstrictor preparations for flexible fibre-optic nasal pharyngoscopy and laryngoscopy. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD005606. doi: 10.1002/14651858.CD005606.pub2. PMID 21412890
- [Background] Miles A, Connor NP, Desai RV, Jadcherla S, Allen J, Brodsky M, Garand KL, Malandraki GA, McCulloch TM, Moss M, Murray J, Pulia M, Riquelme LF, Langmore SE. Dysphagia Care Across the Continuum: A Multidisciplinary Dysphagia Research Society Taskforce Report of Service-Delivery During the COVID-19 Global Pandemic. Dysphagia. 2021 Apr;36(2):170-182. doi: 10.1007/s00455-020-10153-8. Epub 2020 Jul 11. PMID 32654059
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Borrelli B, Sepinwall D, Ernst D, Bellg AJ, Czajkowski S, Breger R, DeFrancesco C, Levesque C, Sharp DL, Ogedegbe G, Resnick B, Orwig D. A new tool to assess treatment fidelity and evaluation of treatment fidelity across 10 years of health behavior research. J Consult Clin Psychol. 2005 Oct;73(5):852-60. doi: 10.1037/0022-006X.73.5.852. PMID 16287385
- [Background] Spillane V, Byrne MC, Byrne M, Leathem CS, O'Malley M, Cupples ME. Monitoring treatment fidelity in a randomized controlled trial of a complex intervention. J Adv Nurs. 2007 Nov;60(3):343-52. doi: 10.1111/j.1365-2648.2007.04386.x. PMID 17908130
- [Background] Honaker J, King, G., Blackwell, M. . Amelia II: A program for missing data. . Journal of Statistical Software 2011;45:1-47.
- [Background] Kutner M, Nachsteim, C., Neter, J., Li, W. . Applied linear statistical models Boston: McGraw-Hill/Irwin; 2005.
- [Background] Schwarz G. Estimating the dimension of a model. The Annals of Statistics 1978;62:461-4.
- [Background] Cameron AC, Windmeijer, F. A. . An R-squared measure of goodness of fit for some common nonlinear regression models. Journal of Econometrics 1997;77:329-42.
- [Background] Lanza ST, Tan X, Bray BC. Latent Class Analysis With Distal Outcomes: A Flexible Model-Based Approach. Struct Equ Modeling. 2013 Jan;20(1):1-26. doi: 10.1080/10705511.2013.742377. PMID 25419096
- [Background] Lanza ST, Rhoades BL. Latent class analysis: an alternative perspective on subgroup analysis in prevention and treatment. Prev Sci. 2013 Apr;14(2):157-68. doi: 10.1007/s11121-011-0201-1. PMID 21318625
- [Background] Lanza ST, Coffman DL, Xu S. Causal Inference in Latent Class Analysis. Struct Equ Modeling. 2013 Jul;20(3):361-383. doi: 10.1080/10705511.2013.797816. PMID 25419097
- [Background] Lanza HI, Huang DY, Murphy DA, Hser YI. A Latent Class Analysis of Maternal Responsiveness and Autonomy-Granting in Early Adolescence: Prediction to Later Adolescent Sexual Risk-Taking. J Early Adolesc. 2013 Apr;33(3):404-428. doi: 10.1177/0272431612445794. PMID 23828712
- [Background] Veterans Affairs Total Parenteral Nutrition Cooperative Study Group. Perioperative total parenteral nutrition in surgical patients. N Engl J Med. 1991 Aug 22;325(8):525-32. doi: 10.1056/NEJM199108223250801. PMID 1906987
- [Background] Pearse RM, Young JD. Steroids to prevent postextubation laryngeal oedema. Lancet. 2007 Mar 31;369(9567):1060-1. doi: 10.1016/S0140-6736(07)60503-0. No abstract available. PMID 17398289
- [Background] Samsoon GL, Young JR. Difficult tracheal intubation: a retrospective study. Anaesthesia. 1987 May;42(5):487-90. doi: 10.1111/j.1365-2044.1987.tb04039.x. PMID 3592174
- [Background] Mallampati SR, Gatt SP, Gugino LD, Desai SP, Waraksa B, Freiberger D, Liu PL. A clinical sign to predict difficult tracheal intubation: a prospective study. Can Anaesth Soc J. 1985 Jul;32(4):429-34. doi: 10.1007/BF03011357. PMID 4027773

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/96/NCT05108896/Prot_SAP_000.pdf